CLINICAL TRIAL: NCT00923897
Title: Phase II Trial of Palliative Radiotherapy for Locally Advanced Hepatocellular Carcinoma and Hepatic Metastases
Brief Title: Palliative Radiotherapy (RT) for Liver Metastases (Mets) and Hepatocellular Carcinoma (HCC)(COLD 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UHN REB 07-0020-CE
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma; Hepatic Metastasis
Keywords: Hepatocellular Carcinoma; Hepatic Metastasis; Palliative Radiation Therapy; Locally advanced HCC and Hepatic Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RT for Liver Mets and HCC (Experimental)
  Interventions: Radiation: Palliative RT

INTERVENTIONS:
Radiation: Palliative RT — Prior to receiving radiation treatment, it is recommended that you take medications to reduce the chance of nausea related to therapy. The treatment will take approximately 30 minutes.

SUMMARY:
Palliative radiotherapy is radiation treatment given to help reduce pain or discomfort, or other symptoms related to cancer. This is used commonly for cancer that has spread to the bones and brain, and for many other primary cancers that are too advanced to be cured, including lung cancer, pancreatic cancer and head and neck cancer. The benefits of palliative radiotherapy for advanced liver cancer have not been well studied.

This study is designed to help to see whether palliative radiation therapy is effective in controlling pain, discomfort or other symptoms related to liver cancer, and how this therapy Phase II Trial of Palliative Radiotherapy for Locally Advanced Hepatocellular Carcinoma and Hepatic Metastases might affect the quality of life of patients receiving such therapy. This information will help the doctors understand if there are specific conditions under which radiation therapy is more effective and worthwhile, and how it may affect the quality of life for patients who have locally advanced hepatocellular carcinoma and hepatic metastasis.

DETAILED DESCRIPTION:
The liver is one of the most common sites with tumour involvement, including both primary and metastatic disease. Gastrointestinal tumours, breast, lung and melanoma are the most common primary sites for hepatic metastases. Hepatocellular carcinoma(HCC) is the sixth most common cancer worldwide, with over 600,000 new cases diagnosed per year. It is the third most common cause of cancer related death.Although, predominately a disease in Asia and sub-Saharan Africa, the incidence of HCC is increasing in North America. The use of radiation in unresectable hepatocellular carcinomas, as well as hepatic metastases, for palliation is uncommon in clinical practice.

This may be because there is a prevailing perception that radiation to the liver will inevitably lead to radiation induced liver disease (RILD). However, several single institution, predominantly retrospective studies, have demonstrated effective palliation for locally advanced HCC as well as hepatic metastases with minimal toxicity.In this study, palliative radiotherapy (RT), delivered in one fraction of 8Gy, will be given to symptomatic patients who are not candidates for radical treatment. We hypothesize that palliative RT will provide symptomatic relief to a large fraction of the patients, with both primary and metastatic disease. We also expect minimal toxicities at this treatment dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma or hepatic metastases from a solid malignancy, unsuitable for radical therapy (including resection, transplant, conformal high dose radiotherapy), confirmed by biopsy or imaging
* Symptoms of hepatic pain, discomfort, nausea, or fatigue requiring palliation
* KPS>60
* Expected survival of greater than 3 months
* Platelet count > 25 bil/L, Hemoglobin > 70 g/L, INR<3, Bilirubin<100 umol/L, AST < 350 U/L or ALT< 400 U/L
* Have signed an informed consent form approved by the Research Ethics Board (REB) at Princess Margaret Hospital

Exclusion Criteria:

* Chemotherapy or novel drug within the past 2 weeks
* TACE(transarterial chemoembolization)within the past 1 month
* Plan for active treatment of the hepatocellular carcinoma or hepatic metastases, including TACE or RFA or ETOH injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
To determine the change in index symptom(s) using an 11 point numerical rating scale for patients with locally advanced hepatocellular cancer or hepatic metastases treated with 8Gy | 5 years

SECONDARY OUTCOMES:
Determine the change in EORTC QLQ-C30 & FACT-Hep for patients with locally advanced HCC/hepatic metastases treated w/h 8Gy and assess the toxicity of treatment using CTC AE v3.0 toxicity score | 5 years
To measure changes in serum cytokines and proteomics following radiotherapy. | 5 years
To determine the feasibility of Cone Beam CT for simulation and treatment and optimize image quality offline. | 5 years
To determine serum marker and radiographic response with 8Gy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Soliman H, Ringash J, Jiang H, Singh K, Kim J, Dinniwell R, Brade A, Wong R, Brierley J, Cummings B, Zimmermann C, Dawson LA. Phase II trial of palliative radiotherapy for hepatocellular carcinoma and liver metastases. J Clin Oncol. 2013 Nov 1;31(31):3980-6. doi: 10.1200/JCO.2013.49.9202. Epub 2013 Sep 23. PMID 24062394